CLINICAL TRIAL: NCT02222337
Title: Nueva Vida Intervention: Improving QOL in Latina Breast Cancer Survivors and Their Caregivers
Brief Title: Nueva Vida Intervention for Latina Breast Cancer Survivors and Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Nueva Vida, Inc. (Industry); Latinas Contra Cancer (Unknown); Gilda's Club NYC (Other); SHARE (Unknown)
Responsible Party: Principal Investigator, Kristi Graves, PhD, Associate Professor, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AD-13-5635
Record Dates: First submitted 2014-08-19; First posted 2014-08-21 (Estimated); Results first posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-02

CONDITIONS: Quality of Life; Breast Cancer
Keywords: behavioral intervention; quality of life; breast cancer; Latina; caregiver; PCORI
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nueva Vida Intervention (Active Comparator): Nueva Vida Intervention consists of 8 sessions of a skills-building group held twice a month for 4 months. Latina survivors and their caregivers arrive at the group together, separate into different rooms to learn the coping and communication skills, and then join together for discussion of the topic.
  Interventions: Behavioral: Nueva Vida Intervention
- Usual Care (No Intervention): Usual care as provided by each of our 4 community-based organization partners. Usual care can include but is not limited to support groups, patient navigation, individual, couple or family therapy.

INTERVENTIONS:
Behavioral: Nueva Vida Intervention — The psycho-educational format of the Nueva Vida Intervention is led by trained interventionists who have the survivors and caregivers go into different rooms to discuss the same topic. This format will allows them each to express their thoughts and feelings without inhibitions or concerns over how their survivor or their caregiver might respond. The specific topics for each wave of the intervention participants will be determined from a larger list of possible topics, with each group including the following core topics: Impact of Cancer on the Family, Spirituality and Cancer, Stress Management, Balancing Physical and Emotional Needs and Improving Communication.
  Arms: Nueva Vida Intervention

SUMMARY:
Latina breast cancer survivors report lower quality of life (QOL) than non-Latina survivors. Lower QOL can lead to poorer functional and cancer-related survival outcomes. The friends and family of Latina cancer patients are also impacted by a loved one's diagnosis of breast cancer. Through strong community-academic partnerships, the investigators seek to improve the QOL of Latina survivors and their caregivers with a culturally-relevant intervention. In this project, the investigators plan to further develop and refine the intervention and then test it through a randomized controlled trial. First, the investigators will conduct in-depth qualitative interviews with 10 survivor-caregiver dyads (pairs) to see if the intervention fits for survivors and caregivers in different parts of the country. Then, the investigators will revise the intervention. Finally, the investigators will test the intervention in a randomized controlled trial. The investigators will invite 125 survivor-caregiver dyads to be a part of our study. Half will be asked to complete the intervention and half will be offered the usual services, such as support groups. The information learned from this study could help improve the quality of life in Latina breast cancer survivors and their caregivers. Physicians, survivors, and community groups can also benefit from this study because they will have more information about the needs of Latina breast cancer survivors. The investigators hope to use the information to help other types of survivors and caregivers in the future.

DETAILED DESCRIPTION:
What is the Nueva Vida Intervention? The "Nueva Vida Intervention: Improving Quality of Life in Latina Breast Cancer Survivors and Their Caregivers" is a randomized controlled trial (RCT) that was co-developed by a Latina breast cancer survivor who is trained as a mental health professional. The program was developed for Nueva Vida, a community-based organization (CBO) in the Washington, DC metropolitan area that serves Latina breast cancer survivors and their families. We are comparing the intervention to the usual services provided at our four partner community-based organizations.

How is the Nueva Vida Intervention Structured? The 8-session psycho-educational quality of life intervention includes group-based skill-building workshops in which Latina survivors and their caregivers are part of concurrently-held but separate groups (survivors in one room; caregivers in another). This separation meets the needs of Latino participants by encouraging them to freely share their experiences and feelings without worrying about upsetting the other person. Five of the eight sessions address core topics: Introduction and The Impact of Cancer on the Family, Stress Management, Improving Communication: Family, Friends, and Providers, Spirituality and Cancer, and Balancing Physical and Emotional Needs.

The remaining three sessions are selected by the intervention participants based on their own needs and interests from the following options: Anger Management, Intimacy after Cancer: Emotional and Sexual, Trauma and Cancer, Role Changes, Understanding Distress and Depression, Myths and Cancer, Including Others in Helping Caregivers, and Putting Our Lives in Order. At the end of the intervention everyone participates in a graduation ceremony.

How does the Nueva Vida Intervention Reflect Latino Values? The Nueva Vida intervention reflects Latino values, including personalismo (warm, personal relationships), familismo (emphasizing the family unit in managing a cancer diagnosis) and framing the sessions as workshops to avoid stigma associated with mental health care.

Where will the Nueva Vida Intervention Study take place? We will evaluate the Nueva Vida Intervention within a multi-site RCT at four community-based organizations in Washington, DC (Nueva Vida), New York, New York (SHARE, Gilda's Club New York City), and San Jose, California (Latinas Contra Cancer).

What is Involved in Study Participation? Latina survivors and their caregivers will be assigned by chance (randomized) to either the Nueva Vida Intervention or to usual care. Survivors and caregivers assigned to usual care can take part in any and all of the services provided at one of the four community-based organizations who are study partners. Both survivors and caregivers will complete informed consent forms and telephone surveys at the beginning of the study, about 4 months later, and again 6 months later. Survivors and caregivers receive gift cards in appreciation of their time for completing the surveys.

ELIGIBILITY:
Inclusion Criteria:

* Survivors: Latina, has been diagnosed with breast cancer, speaks English or Spanish, has a Caregiver who is willing to participate.
* Caregivers: a primary caregiver for a Latina breast cancer survivor, speak English or Spanish

Exclusion Criteria:

1. Inability to understand spoken English and/or Spanish and/or
2. Cognitive impairment that precludes informed consent (determined by the PIs or Co-Investigators who are mental health professionals).

Max Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2013-05; Primary Completion 2017-01-24 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristi D Graves, Ph.D., Principal Investigator — Georgetown University
Locations (4):
- United States (4):
  - Latinas Contra Cancer, San Jose, California
  - Nueva Vida, Washington D.C., District of Columbia
  - Gilda's Club New York City, New York, New York
  - SHARE, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rush CL, Darling M, Elliott MG, Febus-Sampayo I, Kuo C, Munoz J, Duron Y, Torres M, Galvan CC, Gonzalez F, Caicedo L, Napoles A, Jensen RE, Anderson E, Graves KD. Engaging Latina cancer survivors, their caregivers, and community partners in a randomized controlled trial: Nueva Vida intervention. Qual Life Res. 2015 May;24(5):1107-18. doi: 10.1007/s11136-014-0847-9. Epub 2014 Nov 8. PMID 25377349
- See also: Description of the project on the Patient Centered Outcomes Research Institute (PCORI) website — http://www.pcori.org/research-in-action/improving-quality-life-latinas-breast-cancer

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We reconciled the prior enrollment number in the Protocol Section (i.e., "272") that had conflicted with the number of participants started in the Participant Flow module (i.e., "270"). The discrepancy was because two participants enrolled but withdrew prior to the baseline interview. We thus did not have any data on these 2 participants.
Groups:
- Nueva Vida Intervention: Nueva Vida Intervention consists of 8 sessions of a skills-building group held twice a month for 4 months. Latina survivors and their caregivers arrive at the group together, separate into different rooms to learn the coping and communication skills, and then join together for discussion of the topic.
  Nueva Vida Intervention: The psycho-educational format of the Nueva Vida Intervention is led by trained interventionists who have the survivors and caregivers go into different rooms to discuss the same topic. This format will allows them each to express their thoughts and feelings without inhibitions or concerns over how their survivor or their caregiver might respond. The topics for each wave of the intervention participants will be determined from a larger list of possible topics, with each group including the following core topics: Impact of Cancer on the Family, Spirituality and Cancer, Stress Management, Balancing Physical and Emotional Needs and Improving Communication.
Period: Overall Study
Arm/Group | Nueva Vida Intervention | Usual Care
Started | 140 | 132 (132 participants were enrolled but 2 withdrew and never provided any data.)
Completed | 114 | 108
Not Completed | 26 | 24

BASELINE CHARACTERISTICS:
Population: Two participants enrolled in the study but withdrew prior to the baseline interview (thus, N = 130). Baseline analysis was conducted by 1) randomization, and 2) participant type. Data was missing for certain measures; numbers analyzed are adjusted accordingly.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nueva Vida Intervention | Usual Care | Total
Number analyzed (Participants) | 140 | 130 | 270
Age, Categorical [Count of Participants; unit: Participants] — Population: Baseline analysis was conducted by 1) randomization, and 2) participant type. Thus, although there were 140 intervention participants and 130 usual care participants, these groups were separated further to be analyzed by survivor and caregiver status. Further, data was missing for certain measures; numbers analyzed are adjusted accordingly.
  Participants
    Survivors: number analyzed (Participants) | 69 | 65 | 134
    Survivors: <=18 years | 0 | 0 | 0
    Survivors: Between 18 and 65 years | 59 | 56 | 115
    Survivors: >=65 years | 10 | 9 | 19
    Caregivers: number analyzed (Participants) | 67 | 63 | 130
    Caregivers: <=18 years | 0 | 0 | 0
    Caregivers: Between 18 and 65 years | 61 | 57 | 118
    Caregivers: >=65 years | 6 | 6 | 12
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline analysis was conducted by 1) randomization, and 2) participant type. Thus, although there were 140 intervention participants and 130 usual care participants, these groups were separated further to be analyzed by survivor and caregiver status. Further, data was missing for certain measures; numbers analyzed are adjusted accordingly.
  Participants
    Survivors: number analyzed (Participants) | 70 | 65 | 135
    Survivors: Female | 70 | 65 | 135
    Survivors: Male | 0 | 0 | 0
    Caregivers: number analyzed (Participants) | 70 | 65 | 135
    Caregivers: Female | 42 | 38 | 80
    Caregivers: Male | 28 | 27 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Baseline analysis was conducted by 1) randomization, and 2) participant type. Thus, although there were 140 intervention participants and 130 usual care participants, these groups were separated further to be analyzed by survivor and caregiver status. Further, data was missing for certain measures; numbers analyzed are adjusted accordingly.
  Participants
    Survivors: number analyzed (Participants) | 70 | 65 | 135
    Survivors: Hispanic or Latino | 70 | 65 | 135
    Survivors: Not Hispanic or Latino | 0 | 0 | 0
    Survivors: Unknown or Not Reported | 0 | 0 | 0
    Caregivers: number analyzed (Participants) | 70 | 65 | 135
    Caregivers: Hispanic or Latino | 69 | 64 | 133
    Caregivers: Not Hispanic or Latino | 0 | 1 | 1
    Caregivers: Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Baseline analysis was conducted by 1) randomization, and 2) participant type. Thus, although there were 140 intervention participants and 130 usual care participants, these groups were separated further to be analyzed by survivor and caregiver status. Further, data was missing for certain measures; numbers analyzed are adjusted accordingly.
  Participants
    Survivors: number analyzed (Participants) | 70 | 64 | 134
    Survivors: American Indian or Alaska Native | 0 | 0 | 0
    Survivors: Asian | 0 | 0 | 0
    Survivors: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Survivors: Black or African American | 3 | 5 | 8
    Survivors: White | 22 | 17 | 39
    Survivors: More than one race | 28 | 31 | 59
    Survivors: Unknown or Not Reported | 17 | 11 | 28
    Caregivers: number analyzed (Participants) | 70 | 65 | 135
    Caregivers: American Indian or Alaska Native | 0 | 0 | 0
    Caregivers: Asian | 0 | 0 | 0
    Caregivers: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Caregivers: Black or African American | 0 | 1 | 1
    Caregivers: White | 19 | 21 | 40
    Caregivers: More than one race | 25 | 22 | 47
    Caregivers: Unknown or Not Reported | 26 | 21 | 47
Satisfaction with Care Experience of Care and Health Outcomes (ECHOS-NHL) [Mean (Standard Deviation); unit: units on a scale] — This measure was administered to Survivors only. 11 items; Range: 10-44; Higher scores = better communication Population: Baseline analysis was conducted by 1) randomization, and 2) participant type. Thus, although there were 140 intervention participants and 130 usual care participants, these groups were separated further to be analyzed by survivor and caregiver status. Further, data was missing for certain measures; numbers analyzed are adjusted accordingly.
  units on a scale
    number analyzed (Participants) | 69 | 63 | 132
    (all) | 33.68 (5.87) | 34.35 (4.88) | 34 (5.41)
Self-Efficacy - Survivors Only - Cancer Behavior Inventory (CBI) [Mean (Standard Deviation); unit: units on a scale] — 12 items. The CBI-B score is calculated as the sum of all 12 items, range = 12-108. A higher score = higher confidence. Population: Baseline analysis was conducted by 1) randomization, and 2) participant type. Thus, although there were 140 intervention participants and 130 usual care participants, these groups were separated further to be analyzed by survivor and caregiver status. Further, data was missing for certain measures; numbers analyzed are adjusted accordingly.
  units on a scale
    number analyzed (Participants) | 70 | 65 | 135
    (all) | 100.07 (21.28) | 101.60 (19.11) | 100.81 (20.2)
Communication - Patient Satisfaction with Care (PSQ-18 Communication Subscale) [Mean (Standard Deviation); unit: units on a scale] — This scale was administered to Survivors only. 6 items; Range: 1-5; Higher scores = higher general satisfaction with care. Population: Baseline analysis was conducted by 1) randomization, and 2) participant type. Thus, although there were 140 intervention participants and 130 usual care participants, these groups were separated further to be analyzed by survivor and caregiver status. Further, data was missing for certain measures; numbers analyzed are adjusted accordingly.
  units on a scale
    number analyzed (Participants) | 69 | 64 | 133
    (all) | 2.28 (0.91) | 2.28 (0.93) | 2.28 (0.92)
PROMIS Anxiety [Mean (Standard Deviation); unit: units on a scale] — 6 items; Sum and then use IRT to standardize the score. Standardized Mean of 50; SD of 10. Range of the raw score = 6 to 30. Reference value for breast cancer survivors T-score is 49.6. A higher score = higher anxiety. Population: Baseline analysis was conducted by 1) randomization, and 2) participant type. Thus, although there were 140 intervention participants and 130 usual care participants, these groups were separated further to be analyzed by survivor and caregiver status. Further, data was missing for certain measures; numbers analyzed are adjusted accordingly.
  units on a scale
    Survivors: number analyzed (Participants) | 70 | 65 | 135
    Survivors | 54.3 (12.97) | 52.94 (9.95) | 53.65 (11.59)
    Caregivers: number analyzed (Participants) | 70 | 65 | 135
    Caregivers | 51.9 (9.76) | 50.35 (9.26) | 51.15 (9.52)
PROMIS Depression [Mean (Standard Deviation); unit: units on a scale] — 6 items; Sum and then use IRT to standardize the score. Mean of 50; SD of 10. Range of the raw score = 6-30; Reference value for breast cancer survivors T-Score in Depression is 48.5. A higher score = higher depression Population: Baseline analysis was conducted by 1) randomization, and 2) participant type. Thus, although there were 140 intervention participants and 130 usual care participants, these groups were separated further to be analyzed by survivor and caregiver status. Further, data was missing for certain measures; numbers analyzed are adjusted accordingly.
  units on a scale
    Survivors: number analyzed (Participants) | 70 | 65 | 135
    Survivors | 51.35 (12.11) | 48.22 (9.52) | 49.84 (11.01)
    Caregivers: number analyzed (Participants) | 70 | 65 | 135
    Caregivers | 46.72 (9.32) | 45.10 (8.24) | 45.94 (8.82)
PROMIS Fatigue [Mean (Standard Deviation); unit: units on a scale] — 4 items; Sum and then use IRT to standardize the score. Mean of 50; SD of 10. Range of the raw score = 4-20; Reference value for breast cancer survivors T-Score for Fatigue is 52.5. A higher score = higher fatigue Population: Baseline analysis was conducted by 1) randomization, and 2) participant type. Thus, although there were 140 intervention participants and 130 usual care participants, these groups were separated further to be analyzed by survivor and caregiver status. Further, data was missing for certain measures; numbers analyzed are adjusted accordingly.
  units on a scale
    Survivors: number analyzed (Participants) | 68 | 63 | 131
    Survivors | 52.95 (13.03) | 49.57 (11.99) | 51.33 (12.61)
    Caregivers: number analyzed (Participants) | 69 | 65 | 134
    Caregivers | 45.12 (11.24) | 44.14 (9.95) | 44.64 (10.61)
PROMIS Physical Functioning [Mean (Standard Deviation); unit: units on a scale] — 6 items; Sum and then use IRT to standardize the score. Mean of 50; SD of 10. Range of the raw score = 6-28; Reference value for breast cancer survivors T-Score for Physical Functioning is 44.9. A higher score = higher physical functioning Population: Baseline analysis was conducted by 1) randomization, and 2) participant type. Thus, although there were 140 intervention participants and 130 usual care participants, these groups were separated further to be analyzed by survivor and caregiver status. Further, data was missing for certain measures; numbers analyzed are adjusted accordingly.
  units on a scale
    Survivors: number analyzed (Participants) | 70 | 65 | 135
    Survivors | 44.14 (9.15) | 44.33 (9.64) | 44.23 (9.35)
    Caregivers: number analyzed (Participants) | 70 | 65 | 135
    Caregivers | 53.71 (7.54) | 53.72 (7.14) | 53.72 (7.32)
PROMIS Satisfaction With Social Roles [Mean (Standard Deviation); unit: units on a scale] — 6 items; Sum and then use IRT to standardize the score. Mean of 50; SD of 10; Range of the raw score = 6-30; Reference value for breast cancer survivors T-Score for Satisfaction with Social Roles is 50.7. A higher score = higher satisfaction with social roles Population: Baseline analysis was conducted by 1) randomization, and 2) participant type. Thus, although there were 140 intervention participants and 130 usual care participants, these groups were separated further to be analyzed by survivor and caregiver status. Further, data was missing for certain measures; numbers analyzed are adjusted accordingly.
  units on a scale
    Survivors: number analyzed (Participants) | 69 | 63 | 132
    Survivors | 47.79 (7.67) | 48.99 (7.71) | 48.37 (7.68)
    Caregivers: number analyzed (Participants) | 70 | 65 | 135
    Caregivers | 55.18 (8.09) | 55.36 (7.88) | 55.27 (7.96)

OUTCOME MEASURES:

1. Primary Outcome: PROMIS Physical Functioning
Description: Measure Quality of Life physical functioning; 6 items; Sum and then use IRT to standardize the score. Mean of 50; SD of 10. Range of the raw score = 6-28; A higher score = higher physical functioning
Time Frame: 6 months
Population: Cancer survivors
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Usual Care Survivors: Survivors randomized to usual care as provided by each of our 4 community-based organization partners. Usual care can include but is not limited to support groups, patient navigation, individual, couple or family therapy.
- Usual Care Caregivers: Caregivers randomized to usual care as provided by each of our 4 community-based organization partners. Usual care can include but is not limited to support groups, patient navigation, individual, couple or family therapy.
- Nueva Vida Intervetion Survivors: Survivors randomized to the Nueva Vida Intervention: 8 sessions of a skills-building group held twice a month for 4 months. Latina survivors and their caregivers arrive at the group together, separate into different rooms to learn the coping and communication skills, and then join together for discussion of the topic.
  The psycho-educational format of the Nueva Vida Intervention is led by trained interventionists who have the survivors and caregivers go into different rooms to discuss the same topic. This format will allows them each to express their thoughts and feelings without inhibitions or concerns over how their survivor or their caregiver might respond. The topics for each wave of the intervention participants will be determined from a larger list of possible topics, with each group including the following core topics: Impact of Cancer on the Family, Spirituality and Cancer, Stress Management, Balancing Physical and Emotional Needs and Improving Communication.
- Nueva Vida Intervention Caregivers: Caregivers randomized to the Nueva Vida Intervention: 8 sessions of a skills-building group held twice a month for 4 months. Latina survivors and their caregivers arrive at the group together, separate into different rooms to learn the coping and communication skills, and then join together for discussion of the topic.
  The psycho-educational format of the Nueva Vida Intervention is led by trained interventionists who have the survivors and caregivers go into different rooms to discuss the same topic. This format will allows them each to express their thoughts and feelings without inhibitions or concerns over how their survivor or their caregiver might respond. The topics for each wave of the intervention participants will be determined from a larger list of possible topics, with each group including the following core topics: Impact of Cancer on the Family, Spirituality and Cancer, Stress Management, Balancing Physical and Emotional Needs and Improving Communication.
Arm/Group | Usual Care Survivors | Usual Care Caregivers | Nueva Vida Intervetion Survivors | Nueva Vida Intervention Caregivers
Number analyzed (Participants) | 57 | 51 | 57 | 57
units on a scale | 44.61 (8.71) | 53.82 (7.34) | 45.07 (9.20) | 52.99 (7.70)

2. Primary Outcome: PROMIS Satisfaction With Social Roles
Description: Measure Quality of Life satisfaction with social roles domain; 6 items; Sum and then use IRT to standardize the score. Mean of 50; SD of 10; Range of the raw score = 6-30; A higher score = higher satisfaction with social roles
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care Survivors | Usual Care Caregivers | Nueva Vida Intervetion Survivors | Nueva Vida Intervention Caregivers
Number analyzed (Participants) | 57 | 51 | 57 | 57
units on a scale | 52.84 (10.11) | 58.64 (5.93) | 54.07 (9.87) | 59.45 (6.75)

3. Primary Outcome: PROMIS Anxiety
Description: Quality of life: Anxiety; 6 items; Sum and then use IRT to standardize the score. Mean of 50; SD of 10. Range of the raw score = 6 to 30. A higher score = higher anxiety
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care Survivors | Usual Care Caregivers | Nueva Vida Intervetion Survivors | Nueva Vida Intervention Caregivers
Number analyzed (Participants) | 57 | 51 | 57 | 57
units on a scale | 53.93 (12.04) | 48.41 (8.61) | 50.90 (11.99) | 48.70 (8.76)

4. Primary Outcome: PROMIS Depression
Description: Quality of life: depression; 6 items; Sum and then use IRT to standardize the score. Mean of 50; SD of 10. Range of the raw score = 6-30; A higher score = higher depression
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care Survivors | Usual Care Caregivers | Nueva Vida Intervetion Survivors | Nueva Vida Intervention Caregivers
Number analyzed (Participants) | 57 | 51 | 57 | 57
units on a scale | 47.43 (9.46) | 43.95 (7.16) | 47.35 (11.13) | 44.49 (7.48)

5. Primary Outcome: PROMIS Fatigue
Description: Quality of life: fatigue; 4 items; Sum and then use IRT to standardize the score. Mean of 50; SD of 10. Range of the raw score = 4-20; A higher score = higher fatigue
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care Survivors | Usual Care Caregivers | Nueva Vida Intervetion Survivors | Nueva Vida Intervention Caregivers
Number analyzed (Participants) | 57 | 51 | 57 | 57
units on a scale | 49.07 (12.85) | 53.06 (12.38) | 47.83 (10.48) | 46.68 (10.77)

6. Secondary Outcome: Communication - Survivors Only - Patient Satisfaction With Care (PSQ-18 Communication Subscale)
Description: Communication with providers in terms of overall satisfaction with communication. Range for subscale is 1-5; higher scores indicate higher communication satisfaction.
Time Frame: 6-months
Population: Some participants passed away, withdrew, or were lost to follow up after baseline. Data was missing for certain measures; numbers analyzed are adjusted accordingly. Analysis was conducted by 1) randomization, and 2) participant type.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nueva Vida Intervention | Usual Care
Number analyzed (Participants) | 70 | 65
units on a scale | 3.52 (1.94) | 3.23 (1.69)

7. Secondary Outcome: Self-Efficacy - Survivors Only - Cancer Behavior Inventory (CBI)
Description: Self-efficacy; cancer survivors' confidence in coping with cancer and its treatment
Time Frame: 6 Months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nueva Vida Intervention | Usual Care
Number analyzed (Participants) | 70 | 65
units on a scale | 106.96 (19.59) | 107.96 (17.35)

8. Secondary Outcome: Satisfaction With Care - Survivors Only - Experience of Care and Health Outcomes (ECHOS-NHL)
Description: Satisfaction with health care received by the breast cancer survivor from her oncology health care providers or general health care providers
Time Frame: 6-months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nueva Vida Intervention | Usual Care
Number analyzed (Participants) | 70 | 65
units on a scale | 35.04 (4.48) | 34.63 (4.38)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from time of enrollment through 6-month follow-up (3 years).
Arm/Group | Nueva Vida Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 1/140 | 2/130
Serious Adverse Events (participants affected / at risk) | 0/140 | 0/130
Other Adverse Events (participants affected / at risk) | 0/140 | 0/130

LIMITATIONS AND CAVEATS:
Difficulty tracking all approached and eligible participants in terms of number of individuals who declined the study due to recruitment at multiple community events and community sites.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2015-07-08): https://cdn.clinicaltrials.gov/large-docs/37/NCT02222337/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2012-12-17): https://cdn.clinicaltrials.gov/large-docs/37/NCT02222337/Prot_SAP_001.pdf